CLINICAL TRIAL: NCT06362785
Title: Study on the Relationship Between Knee Osteoarthritis, Motor Control and the Risk of Falls, and the Effectiveness of Virtual Reality in Managing It in Older People
Brief Title: Knee Osteoarthritis, Motor Control, Risk of Falls and Virtual Reality
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Collaborators: Centre for Information and Communications Technology Research (CITIC) (Unknown); Faculty of Physiotherapy (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Virtual Reality-Seniors
Record Dates: First submitted 2024-03-26; First posted 2024-04-12 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2024-12

CONDITIONS: Knee Osteoarthritis; Task Performance and Analysis; Accidental Falls; Virtual Reality
Keywords: Knee osteoarthritis; Task Performance and Analysis; Accidental Falls; Aged; Virtual Reality
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- virtual reality (Experimental): The intervention group will perform immersive virtual reality sessions with interactive activities involving functional movements of the spine and limb region in a virtual environment using Meta Quest 3 goggles.
  Interventions: Device: Virtual Reality
- Control (Active Comparator): The control group will receive conventional physiotherapy treatment based on therapeutic exercise.
  Interventions: Behavioral: Therapeutic exercise

INTERVENTIONS:
Device: Virtual Reality — The intervention group will engage in immersive virtual reality sessions with interactive activities involving functional movements of the spine and limbs in a virtual environment using Meta Quest 3 goggles. The intervention will last for 6 weeks, comprising a total of 12 sessions, with a maximum duration of 30 minutes of virtual reality and 15 minutes of rest (45 minutes in total per session).
  Arms: virtual reality
Behavioral: Therapeutic exercise — The control group will receive conventional therapeutic exercise treatment following the recommendations of the Osteoarthritis Research Society International (OARSI), similar to the exercises performed with VR.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn about knee osteoarthritis, functionality, and risk of falls in community-dwelling adults aged 60 years and older. The main questions it aims to answer are:

* What are the characteristics of a community-dwelling population over 60 years and older in terms of knee osteoarthritis, functionality, and risk of falls?
* Does an intervention with virtual reality lower knee osteoarthritis symptoms, raise functionality and prevent falls in community-dwelling adults aged 60 years and older, compared to a control group receiving conventional physiotherapy treatment based on therapeutic exercise?

Participants will:

* Answer questionnaires.
* Perform physical laboratory tests through a camera-based motion capture system.
* Execute task-based exercises in a virtual environment through virtual reality.

Researchers will compare community-dwelling adults aged 60 years and older who execute task based exercises in a virtual environment through virtual reality and community-dwelling adults aged 60 years and older receiving conventional physiotherapy treatment based on therapeutic exercise to see if virtual reality improves knee osteoarthritis symptoms, functionality, and lowers fall risk.

DETAILED DESCRIPTION:
Background

Knee osteoarthritis (OA) is prevalent among older adults, affecting a substantial proportion of this population and being linked to various functional impairments such as joint stiffness, reduced mobility, and chronic pain. More specifically, knee OA is one of the most disabling musculoskeletal conditions worldwide, leading to significant healthcare costs and economic burdens. Several studies have demonstrated a strong association between knee OA and falls in older adults. In particular, it has been observed that knee OA is a significant predictor of multiple falls and is closely related to deficits in balance and gait stability.

To properly understand the close relationship between knee OA and falls, it is crucial to consider motor control dysfunctions associated with joint pain and mechanical alterations, as they are often the primary triggers of falls. Research in this field highlights the importance of directing new studies toward functional tasks, as they represent the essence of motor control. Therefore, the observation and analysis of functional tasks are crucial for examining the motor control of older adults, being 3D motion capture systems the gold standard for the measurement and analysis of human movement.

On the other hand, new technologies such as immersive virtual reality (VR) are gaining recognition and popularity as treatment modalities. This is because they allow users to interact with environments and situations that simulate real life, offering activities tailored to their needs while avoiding the potential risks of the real world. Additionally, it provides an opportunity to repeat exercises, improve performance, and achieve effective learning.

Objectives Several objectives are outlined, as a comprehensive approach involving two different phases will be carried out.

* Phase 1 (Cross-Sectional Study) Main objective: to describe the population aged 60 and older living in the community in terms of knee osteoarthritis symptoms, functionality, and fall risk.
* Phase 2 (Experimental Study) Main objective: to assess the efficacy of a virtual reality intervention in a community-dwelling population aged 60 and above in terms of knee osteoarthritis symptoms improvement, functionality improvement, and fall risk reduction.

Methods

* Setting, locations and relevant dates: testing is going to be conducted in the Research Center for Information and Communication Technologies (CITIC) (A Coruña, Spain) and Senior University Center of the University of A Coruña (A Coruña, Spain).
* Data collection is planned for the months of May 2024 to May 2025.
* Participants: the recruitment of participants will be carried out through the dissemination of the study via informative posters distributed in the University of A Coruña, including the Senior University; in the network of civic centers in the city of A Coruña; as well as electronically through the researchers' social media networks (Twitter, Facebook, and Instagram). The participant information process, as well as the request for informed consent, will be conducted in the CITIC, after having answered the pre-selection questionnaires.
* Variables: see "outcomes measures".
* Study size: the sample size is estimated using the G-power program, indicating that the minimum number of participants needed to detect medium effect sizes, with a type I error probability of 0.05 and a power of 0.95, with an effect size of 0.7 and considering the analysis through the t-test: the difference between two independent means would be a total of 110 participants.
* Statistical analysis: a descriptive analysis will be performed to characterize the subjects in detail. Qualitative variables will be presented as absolute figures with their respective percentages, and quantitative variables as measures of central tendency (mean and median) and dispersion (standard deviation, minimum, and maximum values). The Kolmogorov-Smirnov test will be used to assess the normality of data distribution.

To explore significant differences between groups, a bivariate statistical analysis will be conducted. The Student's T-test for independent samples will be used for comparing means if the variables under consideration are normal; otherwise, the Mann-Whitney U test will be employed for non-normal variables. The chi-square statistic (X2) with a 95% confidence interval will be applied for the association of qualitative variables. The correlation between quantitative variables will be assessed using the Pearson or Spearman correlation coefficient. A significance level of p < 0.05 will be considered. Data processing and analysis will be carried out using the statistical package SPSS, version 24.0 for Windows (Armonk, NY: IBM Corp.).

ELIGIBILITY:
Inclusion Criteria:

* Age over 60 years.
* Non-institutionalized individuals.
* Subjects who wish and consent through informed consent to participate in the study.
* Have the ability to walk independently (with or without assistive devices).
* Diagnosis of primary knee osteoarthritis according to the clinical and radiological criteria of the American College of Rheumatology.
* Specifically, for phase 1, subjects without a knee osteoarthritis diagnosis will also be included.

Exclusion Criteria:

* History of significant previous traumas or surgeries to the spine, pelvis, or legs in the last 12 months.
* Self-reported presence of dizziness, seizures, or epilepsy, aiming to prevent potential exacerbation of symptoms with VR.
* Vestibular disorders (balance).
* Neurological diseases, cardiovascular, or respiratory disorders affecting activity; as well as inflammatory or autoimmune diseases affecting the lower limb joints, and other forms of secondary osteoarthritis.
* Diagnosis of a terminal illness or a health condition that prevents attendance.
* To have a medical contraindication for exercise.
* Body Mass Index (BMI) ≥ 40

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Knee osteoarthritis symptoms | Baseline and change from baseline at 7th week and at 12th month
  Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) is a self-administered questionnaire with 24 items divided into three subscales: (i) pain while walking, using stairs, in bed, sitting, lying down, and standing; (ii) stiffness after waking up and later in the day; (iii) physical function during activities like using stairs, rising from a seated position, bending, walking, getting in/out of a car, shopping, putting on/taking off socks, and performing household tasks. Items are rated on a 0-4 scale: None (0), Mild (1), Moderate (2), Severe (3), Extreme (4). Scores are summed for each subscale (pain: 0-20, stiffness: 0-8, physical function: 0-68). The total score reflects greater pain, stiffness, and functional limitations with higher values.
Pain Intensity | Baseline and change from baseline at 7th week and at 12th month
  Visual Analog Scale (VAS) with a score ranging from 0 to 100 millimeters (mm).
Initial positioning | Baseline and change from baseline at 7th week and at 12th month
  Initial positioning in centimeters (cm) of the spine and limbs through the 3D motion capture system Optitrack, defined as the moment when the orientation angle was 2% greater than the average of the first 20 data points.
Final positioning | Baseline and change from baseline at 7th week and at 12th month
  Final positioning in centimeters (cm) of the spine and limbs through the 3D motion capture system Optitrack, defined as the moment when the orientation angle was 2% lower than the average of the first 20 data points.
Angular velocity | Baseline and change from baseline at 7th week and at 12th month
  Angular velocity of the spine and limbs through the 3D motion capture system Optitrack, determined from the slope of calculated linear regressions for the frames identified from the start to the peak of a movement, measured in degrees per second (°/s).
Acceleration | Baseline and change from baseline at 7th week and at 12th month
  Acceleration of the spine and limbs through the 3D motion capture system Optitrack, defined as the velocity of the spine and limbs change over time in meters per second square (m/s²).
Movement execution time | Baseline and change from baseline at 7th week and at 12th month
  Movement execution time of the spine and limbs through the 3D motion capture system Optitrack, defined as time in seconds to complete or initiate a task.
Range of joint movement | Baseline and change from baseline at 7th week and at 12th month
  Range of joint movement of the spine and limbs through the 3D motion capture system Optitrack, defined as the angle in degrees (°) between the initial and final positions of the spine and limb movements; two 3D vectors defined by the markers to calculate the arctangent.

SECONDARY OUTCOMES:
Kinesiophobia | Baseline
  Tampa Scale for Kinesiophobia (TSK): consists of 11 statements indicating from 1 (completely disagree) to 4 (completely agree) about the fear of movement. A score equal to or greater than 34 indicates kinesiophobia.
Falls history | Baseline and change from baseline at 12th month
  Through an ad hoc question: Have you had any falls in the last year? How many?
General health status | Baseline and change from baseline at 7th week and at 12th month
  Short Form 12 health questionnaire (SF-12): the questionnaire consists of 12 items that assess physical and mental health in eight dimensions. It uses Likert-type scales with 3 to 6 points to measure the intensity and frequency of subjects' health. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
  Additionally, it provides a syntax that compares subjects' scores with reference values for the Spanish population (50±10) in the 8 dimensions and the two summary components (physical and mental) obtained from these dimensions.
Date of birth | Baseline
  Date of birth will be collected as day/month/year.
Gender | Baseline
  Gender will be collected as male or female.
Height | Baseline
  Height of the individual in meters (m) measured using a stadiometer.
Weight | Baseline
  Weight of the individual in kilograms (kg) measured using a scale.
Body mass index (BMI) | Baseline
  Weight and height will be combined to report BMI in kg/m^2.
Depressive symptoms | Baseline and change from baseline at 7th week and at 12th month
  Through the Geriatric Depression Scale (GDS-15), which consists of 15 questions with 2 response options (yes/no). The scale's scoring includes: 0-5: normal; >5: depression.
Cognitive capacity | Baseline and change from baseline at 7th week and at 12th month
  Trail Making Test (TMT), which consists of two parts (A and B). It involves connecting letters and numbers as quickly as possible without making mistakes. In Part A, the cutoff point between normal and impaired attention is 75 seconds. In Part B, the cutoff point between normal executive function and impairment is >180 seconds. The test is considered complete when Part A exceeds 100 seconds and Part B exceeds 300.
Amount and type of medication consumed | Baseline and change from baseline at 7th week and at 12th month
  Through an ad hoc question: In case of taking medication, what type of medication do you use? How often per day/week?
Existence of comorbidity | Baseline
  Through the Charlson Comorbidity Index. The score on this index includes: 0-1 point: absence of comorbidity; 2 points: low comorbidity; >3 points: high comorbidity.
Physical performance and fall risk | Baseline and change from baseline at 7th week and at 12th month
  4x10 m Fast-Paced Walk Test: This test measures the total time (in seconds) required to walk a 10-meter distance four times as fast as possible without running. Times below 8 seconds indicate excellent functional mobility, times between 8 and 12 seconds reflect adequate mobility with slight limitations, and times exceeding 12 seconds suggest significant functional impairment.
Lower limb strength and function | Baseline and change from baseline at 7th week and at 12th month
  Stair Climb Test: This test measures the time (in seconds) it takes for a person to ascend and descend a predefined number of steps. Times below 10 seconds indicate good functional capacity, times between 10 and 15 seconds are considered acceptable, while times exceeding 15 seconds suggest reduced functional capacity and possible muscle weakness.
Mobility and balance | Baseline and change from baseline at 7th week and at 12th month
  Timed Up and Go (TUG) Test: This test measures the time (in seconds) required to stand up from a chair, walk 3 meters, turn around, and return to the chair to sit down again. A result below 10 seconds represents excellent mobility, times between 11 and 20 seconds are considered normal, and times exceeding 20 seconds indicate mobility limitations and a higher risk of falls.
Muscle Strength | Baseline and change from baseline at 7th week and at 12th month
  30-Second Chair Stand Test: This test measures the number of times a person can stand up from and sit down on a chair within 30 seconds. More than 14 repetitions indicate adequate lower limb muscle strength, between 8 and 14 repetitions reflect moderate strength with potential for improvement, and fewer than 8 repetitions suggest muscle weakness and possible functional limitations.
Aerobic capacity | Baseline and change from baseline at 7th week and at 12th month
  6 Minutes Walking Test (6MWT): this test measures the total distance covered in 6 minutes at a self-paced speed. Walking more than 500 meters indicates excellent functional capacity, between 400 and 500 meters reflects normal capacity with a slight decline, while distances under 400 meters signal significant physical endurance limitations.
Heart Rate | Baseline and change from baseline at 7th week and at 12th month
  HR: Measured using a pulse oximeter or smartwatches/fitness trackers. At rest, normal values range from 50 to 100 beats per minute (bpm). A rate over 100 bpm may indicate stress or cardiovascular issues, while values below 50 bpm may reflect good physical conditioning.
Blood Pressure | Baseline and change from baseline at 7th week and at 12th month
  BP: Measured using a sphygmomanometer. Normal values are below 120/80 mmHg. Values between 120/80 and 139/89 mmHg indicate prehypertension, while readings above 140/90 mmHg suggest hypertension and an increased cardiovascular risk.
Oxygen Saturation | Baseline and change from baseline at 7th week and at 12th month
  SpO2: Measured using a pulse oximeter. Normal values range from 95% to 100%. Values below this range may indicate insufficient oxygen levels.
Cibersickness | Baseline and change from baseline at 7th week and at 12th month
  Simulator Sickness Questionnaire (SSQ): assesses symptoms associated with VR use through three subscales (nausea, disorientation, and fatigue) and a total score. A score of 0-20 points reflects a low level of symptoms and adequate tolerance; 21-40 indicates moderate symptoms with mild discomfort; 41-100 points signify a high level of symptoms with noticeable discomfort; and values above 100 represent severe discomfort, requiring an immediate interruption of VR use.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Rodríguez-Romero, PhD, Study Director — Universidade da Coruña

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be openly available in Zenodo.
Supporting Information: CSR
Time Frame: The supporting information will be available in the official repository of the University of A Coruña for an indefinite period of time.
Access Criteria: Upon request of access to the authors of the study.
URL: https://www.udc.es/es/biblioteca.fic/recursos_informacion/repositorios/

REFERENCES:
- [Background] Altenburger P, Ambike SS, Haddad JM. Integrating Motor Variability Evaluation Into Movement System Assessment. Phys Ther. 2023 Oct 3;103(10):pzad075. doi: 10.1093/ptj/pzad075. PMID 37364059
- [Background] Quinn L, Riley N, Tyrell CM, Judd DL, Gill-Body KM, Hedman LD, Packel A, Brown DA, Nabar N, Scheets P. A Framework for Movement Analysis of Tasks: Recommendations From the Academy of Neurologic Physical Therapy's Movement System Task Force. Phys Ther. 2021 Sep 1;101(9):pzab154. doi: 10.1093/ptj/pzab154. PMID 34160044
- [Background] Benham S, Kang M, Grampurohit N. Immersive Virtual Reality for the Management of Pain in Community-Dwelling Older Adults. OTJR (Thorofare N J). 2019 Apr;39(2):90-96. doi: 10.1177/1539449218817291. Epub 2018 Dec 29. PMID 30595096
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Stratford PW, Kennedy DM, Woodhouse LJ. Performance measures provide assessments of pain and function in people with advanced osteoarthritis of the hip or knee. Phys Ther. 2006 Nov;86(11):1489-96. doi: 10.2522/ptj.20060002. PMID 17079748
- [Derived] Tunas-Maceiras I, Pereira J, Pertega Diaz S, Lopez Campos JA, Rodriguez-Romero B. Virtual reality versus conventional exercise for knee osteoarthritis: protocol for a randomised controlled trial on functionality and fall risk. BMJ Open. 2025 Oct 20;15(10):e102776. doi: 10.1136/bmjopen-2025-102776. PMID 41120141